CLINICAL TRIAL: NCT05039528
Title: Design and Usability Testing of a Tailored Intervention to Increase Awareness About Sleep and Sleep Disorders Among Transportation Workers
Brief Title: Design and Usability Testing of a Tailored Intervention About Sleep and Sleep Disorders Among Transportation Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rebecca Robbins, Assistant Professor of Medicine at Harvard Medical Scool and Associate Scientist at Brigham & Women's Hospital, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019P003171; K01HL150339 (NIH)
Record Dates: First submitted 2021-07-12; First posted 2021-09-09 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: A 2-month pre-post pilot study will be conducted. Two worksites will be selected at random then randomized to either the tailored (intervention) or non-tailored (control) groups. Participants who fit the eligibility criteria will be recruited from each worksite and assigned to the study arm corresponding to their worksite (20 per worksite for a total of 40 participants).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive the personalized OSA messages.
  Interventions: Behavioral: Personalized OSA messages
- Control (Placebo Comparator): Placebo participants will receive no treatment during the experiment.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Personalized OSA messages — Participants will receive personalized OSA messages designed to nudge and navigate them toward evaluation and treatment for OSA. Participants will complete questionnaires at baseline and at study follow-up.
  Arms: Intervention
Other: Control — Participants will complete questionnaires at baseline and at study follow-up. At the end of the study period, participants will receive the OSA message intervention.
  Arms: Control

SUMMARY:
The objective of this protocol is to conduct a focus group to identify OSA beliefs, attitudes, and knowledge among employees in the transportation industry on shift schedules.

DETAILED DESCRIPTION:
Transportation shift workers (TSW, e.g., overnight, on-call, or rotating) have been identified as a high-risk group for health conditions (e.g., obesity, cardiovascular disease). Also, TSW are at risk for obstructive sleep apnea (OSA). According to one study, approximately 36% of TSWs have OSA, a condition that exacerbates health risks and daytime sleepiness. A recent report from the American Academy of Sleep Medicine (AASM) showed that those with untreated OSA cost on average $4,261 more than those without OSA. Also concerning, workers with OSA who are non-adherent to recommended OSA treatment (i.e., continuous positive airway pressure, CPAP) are at particularly high risk for motor vehicle accidents compared to those who are adherent.

This protocol outlines focus groups that will aim to identify knowledge, attitudes, and beliefs about OSA among TSW. Results of these focus groups will be used in future research to design a tailored website for relaying OSA information to TSW.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Access to a smartphone device
3. Commitment to completing all study activities
4. Score 4 or higher (mild or higher on OSA risk) according to the Apnea Risk Evaluation System (ARES) questionnaire.

Exclusion Criteria:

1. Significant medical or psychiatric illness according to the PROMIS Short Form (SF-12)
2. No OSA risk (a score below 4 on the ARES).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change in OSA self-management efficacy as measured by the Survey of OSA Functional Health Literacy (SOFHL) | The SOFHL will be administered at baseline and post-intervention. Change in SOFHL score on self-management efficacy will be computed by comparing responses at baseline and post-intervention.
  OSA self-management efficacy will be examined using the SOFHL

SECONDARY OUTCOMES:
Change in OSA general knowledge as measured by the SOFHL. | The SOFHL will be administered at baseline and post-intervention. Change in SOFHL score on OSA general knowledge will be computed by comparing responses at baseline and post-intervention.
  OSA general knowledge will be assessed with the validated SOFHL.
Change in Daytime sleepiness as measured by the Epworth Sleepiness Scale (ESS). | Sleepiness will be assessed at baseline and post-intervention. Change in daytime sleepiness will be computed by comparing responses at baseline and post-intervention..
  Daytime sleepiness will be assessed with the validated ESS.
Change in Attentional Failures as measured by previously validated questions assessing Attentional Failures. | Attentional failures will be measured at baseline and post-intervention.Change in attentional failures will be computed by comparing responses at baseline and follow-up.
  Attentional failures (e.g., near miss accidents) will be measured via self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Robbins, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No